CLINICAL TRIAL: NCT04822532
Title: Implementing Pharmacogenetics in the Busulfan Dosing Method for Children Undergoing Hematopoietic Stem-cell Transplantation: a Prospective, Multicentric, Randomized Clinical Trial
Brief Title: Precision Dosing of Busulfan in Children Undergoing HSCT
Acronym: BuGenes01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Marc Ansari, Professeur Marc Ansari, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BuGenes 01
Record Dates: First submitted 2021-03-12; First posted 2021-03-30 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-03

CONDITIONS: Hematopoietic Stem Cell Transplantation; Allogeneic Hematopoietic Stem Cell Transplantation; Autologous Hematopoietic Stem Cell Transplantation
Keywords: Precision dosing; Pharmacogenetics; Children; Adolescent; Busulfan; HSCT

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacogenetic based-model (GSTA1) (Experimental)
  Interventions: Genetic: GSTA1 genotyping
- The most performing method based on age and weight - McCune's model (Active Comparator)
  Interventions: Genetic: GSTA1 genotyping

INTERVENTIONS:
Genetic: GSTA1 genotyping — Diplotype determination based on 4 single-nucleotide polymorphisms (SNPs) occurring in the promoter region of the GSTA1 gene

SUMMARY:
The objective of this clinical trial is to evaluate the personalization the conditioning regimen prior to the hematopoietic stem cell transplant (HSCT) in children and adolescents, to improve HSCT efficacy while reducing conditioning-related toxicities. Namely, we are going to compare the accuracy of two methods for determining the first dose of busulfan, one of the medicines used during the conditioning regimen. First doses will be determined based either only on anthropometric information such as age and weight or by adding a genetic factor that influences the individual ability of busulfan metabolization.

DETAILED DESCRIPTION:
Participants will be randomly assigned (1:1 ratio, stratified by conditioning regimen - the presence of fludarabine) to receive their first dose of busulfan according to:

1. the most performing method based on age and weight - McCune's model (control arm)
2. a method that also considers a pharmacogenetic factor (variants occurring in the promoter region of the GSTA1 gene) in association with the co-administered chemotherapeutic agent fludarabine in the dose personalization (experimental arm)

This is an international study being carried out in five countries (Canada, Italy, Switzerland, France, and Denmark).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be aged from 0-18 years old on entry to the study;
* Clinical indication of allogeneic or autologous hematopoietic stem cell transplantation;
* The conditioning protocol must include IV Bu formulations, Busulfex® (Otsuka Pharmaceutical), Busilvex® (Pierre Fabre Pharma) or other European Medicines Agency (EMA) or Food and Drugs Administration (FDA) approved generic formulations regardless of the administration schedule (q6h, q12h, or q24h)
* The expected length of time from recruitment to starting the conditioning regimen must be superior to 10 days;
* Informed written consent to participate in the study signed by the participant/parent

Exclusion Criteria:

• At least one of the drugs listed below scheduled to be administered in the Bu administration days up to 24h after the last dose of Bu, whenever a washout is not possible:

* Metronidazol (required washout: 7 days)
* Nalidixic acid (required washout: 7 days)
* Phenytoin (required washout: 21 days)
* Itraconazole (required washout: 14 days)
* Ketoconazole (required washout: 7 days)
* Voriconazole (required washout: 7 days)
* Deferasirox (required washout: 7 days)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the first-dose Bu area under the curve (AUC) prediction | 1 month
  Proportion of the first doses which result in AUCs within the therapeutic target range defined by the prescriber
Accuracy of the Bu Clearance prediction | 1 month
  Absolute prediction error between the predicted and measured Bu clearance of the first dose
Dose adjustment requirement | 1 month
  Change in percentage between the first dose administered and the next time-wise adjustable dose: 2nd (Bu q24h), 3rd (Bu q12h), or 5th (Bu q6h) doses

SECONDARY OUTCOMES:
Time to deliver the personalized dose | 1 week
  Proportion of personalized doses delivered within the optimal delivery time (to be determined during the first year of the trial)
Incidence of treatment-related toxicities (TRTs) | 12 months
Incidence and severity of sinusoidal obstruction syndrome (SOS) | 12 months
Incidence of primary and secondary graft failure | 12 months
Incidence and severity of acute graft-versus-host disease (aGVHD) | 12 months
Overall survival | 12 months
Event-free survival | 12 months
  Considering as event aGVHD, SOS, relapse and death

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCune JS, Bemer MJ, Barrett JS, Scott Baker K, Gamis AS, Holford NH. Busulfan in infant to adult hematopoietic cell transplant recipients: a population pharmacokinetic model for initial and Bayesian dose personalization. Clin Cancer Res. 2014 Feb 1;20(3):754-63. doi: 10.1158/1078-0432.CCR-13-1960. Epub 2013 Nov 11. PMID 24218510
- [Background] Nava T, Kassir N, Rezgui MA, Uppugunduri CRS, Huezo-Diaz Curtis P, Duval M, Theoret Y, Daudt LE, Litalien C, Ansari M, Krajinovic M, Bittencourt H. Incorporation of GSTA1 genetic variations into a population pharmacokinetic model for IV busulfan in paediatric hematopoietic stem cell transplantation. Br J Clin Pharmacol. 2018 Jul;84(7):1494-1504. doi: 10.1111/bcp.13566. Epub 2018 Apr 27. PMID 29469189
- [Background] Hassine KB, Nava T et al. 2021 (manuscript submitted).